CLINICAL TRIAL: NCT02872298
Title: A pRospective, Multicenter, Single-arm Study EvaLuating the Safety and feasIbility of Targeted Lung Denervation (TLD) for the trEatment oF Severe Asthma
Brief Title: Evaluating the Safety and Feasibility of TLD for the Treatment of Severe Asthma
Acronym: RELIEF-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Nuvaira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0384
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Asthma
Keywords: Severe; Refractory
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment: Targeted Lung Denervation (TLD)
  Interventions: Device: Targeted Lung Denervation (TLD)

INTERVENTIONS:
Device: Targeted Lung Denervation (TLD) — The Nuvaira Lung Denervation System, manufactured by Nuvaira, Inc., is intended to deliver TLD Therapy using predetermined radiofrequency (RF) energy over a predetermined period of time to ablate airway nerve trunks which are located on the outside of the main bronchi.

SUMMARY:
Prospective, multicenter, single-arm (non-randomized) study of Targeted Lung Denervation (TLD) Therapy in subjects with severe asthma.

DETAILED DESCRIPTION:
Prospective, multicenter, single-arm (non-randomized) study. All patients will undergo a run in period on optimal medical therapy as part of eligibility testing. Final determination to initiate treatment will be made after initial airway inspection. A total of 20 patients will be treated. Inflammatory biomarkers (washes and brushes) will be collected in all patients and bronchial biopsies will be collected from the last 10 patients at the time of treatment and at 90-days post-treatment. All patients will be prescribed peri-procedural antibiotics and steroids to minimize procedural risks. All patients will be provided a mobile handheld spirometer to measure and record daily peak expiratory flow both before and after treatment to monitor lung function. Patient follow-up will be conducted out to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent;
* Diagnosis of severe asthma as defined by the 2018 GINA Report, and are taking regular maintenance medication as specified in the study protocol;
* Pre-bronchodilator FEV1 ≥50% predicted after a 4 week medication run-in;
* Subject has at least two days of asthma symptoms during the 4-weeks of the Baseline Diary Period;
* Women of child bearing potential must have a negative pregnancy test and agree not to become pregnant for the duration during the study;
* Non-smoker for at least 6 months and agree to continue not smoking for duration of the study;
* Patient is a candidate for bronchoscopy in the opinion of the physician or per hospital guidelines;
* Patient is a candidate to undergo methacholine challenge testing;
* Patient is willing, able and agrees to complete all protocol required baseline and follow up testing and comply with medication requirements.

Exclusion Criteria:

* In the 24 months prior to enrollment, the subject has: been intubated for asthma, had intensive care unit (ICU) admission(s) for asthma, or been treated with immunosuppressant therapy for any reason (steroids excluded);
* In the 12 months prior to enrollment, the subject has had: ≥4 lower respiratory tract infections requiring antibiotics or ≥4 hospitalizations for asthma exacerbations;
* In the 3 months prior to enrollment, the subject has taken/used an opioid(s);
* In the 6 weeks prior to enrollment the subject has had a lower respiratory tract infection or asthma exacerbation that required: antibiotics, unscheduled physician visits for asthma care, changes in use of asthma maintenance medication, taking of rescue medication over normal dose in a 24-hour period for asthma symptoms and a steroid burst (pulse);
* Current use of greater than 10 mg of oral steroids per day at the time of enrollment;
* History of poor medication compliance;
* Prior lung or chest procedure;
* Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal chord dysfunction, eosinophilic granulomatosis with polyangiitis (EGPA) or interstitial lung disease that is the sole cause of asthma symptoms, severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways;
* Pre-existing diagnosis of pulmonary hypertension as defined in the study protocol;
* Uncontrolled diabetes as evidenced by an HbA1c > 7%;
* Patient has an implantable electronic device;
* Known contraindication or allergy to anticholinergic drugs or components;
* Known contraindication of allergy to medications required for bronchoscopy, general anesthesia or peri-procedural therapy that cannot be medically controlled;
* Patient is unable to stop blood thinning medication for 7 days prior and 7 days after procedure;
* Documented history of untreated severe obstructive sleep apnea;
* Patient has any disease or condition that might interfere with completion of a procedure or this study or patient safety;
* Screening chest CT scan reveals bronchi anatomy cannot be fully treated with the available catheter sizes or discovery of a pulmonary nodule requiring follow-up or intervention unless proven benign;
* Patients who had abdominal surgical procedures on stomach, esophagus or pancreas;
* Patients with a Gastroparesis Cardinal Symptom Index (GCSI) score ≥ 18 prior to treatment;
* Patient is currently enrolled in another clinical trial that has not completed follow-up.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Freedom from device related therapeutic interventions | 7 days, 1 month, 3 months, 6 months, and 12 months post-procedure
  Number and % of patients free from device related therapeutic interventions will be reported. Therapeutic intervention is defined as administration of non-protocol required antibiotics or steroids, an endoscopic procedure or surgery to treat findings and/or conduction of another diagnostic test to assess the treatment area due to safety concerns.

SECONDARY OUTCOMES:
Device Success | 1 day
  Number and % of subjects with reported Device Success, defined as the ability to insert and place the dNerva Catheter to its intended locations and intact removal.
Technical Success | 1 day
  Number and % of subjects with reported Technical Success, defined as device success with the ability to deliver RF energy to each intended location as confirmed by the Nuvaira Console.
Change in Quality of Life (QOL) | Through study completion, an average of 3 years
  Changes in the Asthma Quality of Life Questionnaire (AQLQ) over time will be assessed. Comparisons will be made to baseline score.
Change in Asthma Control | Through study completion, an average of 3 years
  Changes in the Asthma Control Questionnaire (ACQ) over time will be assessed. Comparisons will be made to baseline score.

OTHER OUTCOMES:
Rate of respiratory and non-respiratory adverse events | Through study completion, an average of 3 years
  Rate of respiratory and non-respiratory adverse events
Change in morning and evening peak expiratory flow (PEF) | Through 1 year follow-up
  Change in morning and evening peak expiratory flow (PEF)
Change in pre- and post-bronchodilator FEV1 | Through study completion, an average of 3 years
  Change in pre- and post-bronchodilator FEV1 at pre-specified time points from baseline.
Change in methacholine PC20 | Through 1 year follow-up
  Change in methacholine PC20 (provocation concentration causing a 20% fall in FEV1) at pre-specified time points from baseline.
Change in rescue medication usage | Through study completion, an average of 3 years
  Change in rescue ("reliever") medication usage
Number and level of asthma exacerbations | Through study completion, an average of 3 years
  Number and level of asthma exacerbations
Number of respiratory-related unscheduled physician office visits | Through study completion, an average of 3 years
  Number of respiratory-related unscheduled physician office visits
Number of emergency department visits | Through study completion, an average of 3 years
  Number of emergency department visits
Number of hospitalizations | Through study completion, an average of 3 years
  Number of hospitalizations
Change in inflammatory markers and bronchoscopic specimens | 90 days
  Analysis of inflammatory markers and bronchoscopic specimens collected at treatment and 90 days post-treatment.
Change in visual and quantitative lung attenuation via CT scan | 1 Year
  CT assessment includes visual and quantitative lung attenuation statistics and texture analyses, airway morphometry, regional airflow and airway reactivity, air trapping and structural changes.
Change in Cough | Through study completion, an average of 3 years
  Changes in the Leicester Cough Questionnaire (LCQ) over time will be assessed. Comparisons will be made to baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Nick ten Hacken, MD, Principal Investigator — University Medical Center Groningen (UMCG); Pallav Shah, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (9):
- CHU de Grenoble, Grenoble, France
- Thoraxklinik Heidelberg, Heidelberg, Germany
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Universtity Medical Center Groningen, Groningen
- United Kingdom (5):
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Chelsea & Westminster Hospital NHS Foundation Trust, London
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - NUH Nottingham City Hospital, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No